CLINICAL TRIAL: NCT01570959
Title: A Two Period, Two Treatment, Two Way, Steady State Crossover Bioequivalence Study of Quetiapine Fumarate 300 mg Tablets Under Fasting Conditions
Brief Title: Crossover Bioequivalence Study of Quetiapine Fumarate 300 mg Tablets Under Steady State Fasted Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Sponsor
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: QUET-T300-PVSS
Record Dates: First submitted 2012-03-28; First posted 2012-04-04 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Bipolar I Disorder
MeSH Terms: interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Quetiapine Fumarate — 300 mg tablet
  Other Names: Seroquel

SUMMARY:
The objective of this study was to prove the bioequivalence of Roxane Laboratories' Quetiapine Fumarate 300 mg Tablet under fasted steady state conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Stable patients with the DSM-IV TR diagnosis of schizophrenia. These patients are to be identified via psychiatric evaluation and meet DSM-IV TR criteria for schizophrenia of paranoid (295.30), disorganized (295.10), catatonic (295.20), undifferentiated (295.90), or residual (295.60) subtype.
2. Patient to have no significant breakthrough symptoms or exacerbations of psychiatric illness necessitating hospitalization in the 3 months prior to screening.
3. Patient to have a CGI-S score of 3 or less at screening.
4. On a stable regimen of treatment to include quetiapine fumarate for 3 months minimum prior to screening, and on a dose of quetiapine fumarate totaling 600 mg total per day for a minimum of 1 month prior to screening. Patients who are on qd dosing of daily quetiapine fumarate must be willing to convert to 300 mg bid dosing for the duration of the study.

Exclusion Criteria:

1. All other DSM-IV axis I diagnoses, including schizoaffective disorder, schizophreniform disorder and/or any other psychiatric diagnoses that in the opinion of the principal investigator may during the conduct of the trial become a primary treatment concern, or may interfere in the patients ability to participate in the trial.
2. Positive test for HIV, Hepatitis B, or Hepatitis C.
3. Treatment with known enzyme altering drugs.
4. History of allergic or adverse response to quetiapine or any comparable or similar product.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2007-04; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
bioequivalence determined by statistical comparison Cmax | 10 days

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - Synergy Clinical Research Center, National City, California
  - Segal Institute for Clinical Research, North Miami, Florida
  - Global Medical Institutes/Princeton Medical Institute, Princeton, New Jersey
  - CRI Worldwide, Willingboro, New Jersey
  - Community Clinical Research, Inc., Austin, Texas
  - Claghorn-Lesem Research Clinic, Ltd, Houston, Texas